CLINICAL TRIAL: NCT04978896
Title: Can a Self-guided Program on a Mobile Application Improve Wellbeing and Stress Coping? - A Randomized Controlled Trial
Brief Title: Effectiveness of a Self-guided Mobile Application in Improving Wellbeing and Stress Coping
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: Intellect Pte. Ltd. (Industry)
Responsible Party: Principal Investigator, Dr Oliver Suendermann, Deputy Director Master in Clinical Psychology Program, National University of Singapore
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: NUS-IRB-2021-242
Record Dates: First submitted 2021-07-18; First posted 2021-07-27 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Stress

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group: Stress-coping Program (Experimental): Participants will complete an 8-day self-guided programme on stress-coping delivered via a mobile-phone application with daily exercises guided by cognitive-behavioural principles.
  Interventions: Device: Self-guided program on stress coping
- Control group (Active Comparator): Participants will complete an 8-day self-guided programme on cooperation delivered via a mobile-phone application with daily exercises that differ to the intervention group in terms of content but are comparable in terms of duration.
  Interventions: Device: Self-guided program on cooperation

INTERVENTIONS:
Device: Self-guided program on stress coping — This is an 8-day program that provides psychoeducation on the negative effects of stress and effective stress-management skills to combat stress. Guided by principles of CBT, the program targets the thoughts and behaviours of participants and equips them with skills to alter negative cognitions pertaining to stress. Participants are engaging with a series of exercises involving reflection and mindfulness where they are required to spot and write down their stressors, the negative thoughts associated with the stressors, as well as positive affirmations. Participants will also be taught breathing exercises and are encouraged to practice them during 2 check-ins.
  Arms: Intervention group: Stress-coping Program
Device: Self-guided program on cooperation — The 8-day program on cooperation aims to provide psychoeducation for participants to understand and improve collaboration and interpersonal relationships. Short quizzes and practice exercises on feedback-giving will be included. The time and duration of the cooperation SGA is matched to the stress-coping SGA to ensure that participants spend a similar amount of time and effort across both the intervention and active-control conditions.
  Arms: Control group

SUMMARY:
Excessive and chronic stress is a major public global health concern. Young adults are at particular risk to experience heightened stress because of life transitions. Short skills-focused self-guided applications (SGA) on mobile phones are a cost-effective and scalable way to equip users with better stress-coping skills, but many SGA stress-coping programmes are not evidence-based, existing research is flawed with methodological problems and is also predominantly conducted in Western countries. Questions also remain for whom SGAs work (moderators) and by which pathways (mediators).

This study is a randomised-controlled trial (RCT) that evaluates the effectiveness of a recently developed mobile-phone SGA in improving stress coping in young adults.

Hypothesis 1: The intervention group will report significantly lower stress symptoms at post-intervention and 1-month follow-up compared to the control group.

Hypothesis 2: Coping self-efficacy will mediate the expected relationship between the use of the Stress-SGA and lower stress symptoms, i.e. people with higher coping self-efficacy will benefit more from the Stress-SGA than those with lower coping self-efficacy.

Hypothesis 3: Psychological mindedness will moderate the expected relationship between the use of Stress-SGA and lower stress symptoms, i.e. people high in psychological mindedness will benefit more from the Stress-SGA than those with lower psychological mindedness.

DETAILED DESCRIPTION:
Procedure:

Participants will sign up for the study via a survey link posted on the university's recruitment sites, where they will first read through the Participant Information Sheet, which contains information about the study such as study aims, methods, benefits and risks, the confidentiality of data, and contact information of the investigators. If participants agree to participate, they will provide their consent on the online consent form. Thereafter, they will proceed to complete a series of self-report measures on an online survey platform (baseline ratings). The online survey consists of the primary outcome measures on stress (PSM-9, PHQ-9 & GAD7), secondary outcome measures on coping self-efficacy and psychological mindedness (CSES & PM), and demographic information (age, gender).

Next, participants will be randomly assigned to either the intervention or active control condition and guided to download the SGA on their personal mobile devices from the Apple App Store or Google Play Store. A number code will be provided to them to unlock the app according to their assigned condition. The SGA is developed by Intellect Pte Ltd, a Singapore based technology firm that collaborates with the supervisor of the study. Participants in the intervention condition will take part in the 8-day stress management program while those in the active control condition will take part in the 8-day cooperation learning program. Both programs will involve content education and short daily activities, averaging about five minutes, to fulfil a series of tasks aimed at improving their wellbeing. Daily reminders to complete the program will be sent via text messages by the researcher to participants. All participants will be instructed to refrain from engaging in any self-guided wellbeing apps other than the given SGA during the duration of the study, lasting from the beginning until the end of the 1-month follow-up. This minimises potential confounding effects.

Upon completion of the 8-day program, participants will receive a survey link to complete the same questionnaires and in addition, will fill out the App Engagement Scale. One month upon completion of the SGA, participants will be emailed the survey link to the self-report measures again, along with the debrief and an information sheet explaining the main purposes of the study. All participants will be given a link to access the complete version of the SGA, providing them with access to all the wellbeing programs available for their personal use. Participants will be reimbursed with either course credit or a small monetary fee for their time and effort..

ELIGIBILITY:
Inclusion Criteria:

* Age 18-30
* Good command of the English Language

Exclusion Criteria:

* None

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 323 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Change of psychological stress | Baseline, 8 days (completion of intervention), 4 weeks (follow-up)
  Psychological Stress Measure (PSM-9; Lemyre & Tessier, 1988) is used to measure the affective, cognitive, behavioural, and somatic components of psychological stress. This is a 9-item self-report measure utilising a 8-point scale (1 = 'Not at all', 8 = 'Extremely'). Some examples of the items include "I feel calm" and "I feel a great weight on my shoulders". Low ratings on items 1 and 6 and high ratings on the other items demonstrate greater symptomatology. When calculating for the total score, the opposite value of the rating will be given to items 1 and 6, where a rating of 1 = 8 points and conversely, a rating of 8 = 1 point. This results in higher total scores reflecting more stress symptoms. The PSM-9 is found to have excellent internal consistency where Cronbach׳s α = .89.

SECONDARY OUTCOMES:
Change in depressive symptoms | Baseline, 8 days (completion of intervention), 4 weeks (follow-up)
  The Patient Health Questionnaire (PHQ-9; Kroenke et al., 2001) is a widely-used 9-item measure of depression symptoms. Stress symptoms often include low mood and depression, rendering the measuring of depression symptoms to be valid in identifying stress levels. Items include "Feeling down, depressed, or hopeless" and "Poor appetite or overeating". Items are scored on a 4-point scale (0 ='Not at all'; 3 = 'Nearly every day'). It has been found to have an excellent internal consistency of Cronbach's α=0.89.
Change in generalised anxiety | Baseline, 8 days (completion of intervention), 4 weeks (follow-up)
  Generalised Anxiety Disorder scale (GAD-7; Spitzer et al., 2006) is a 7-item self-report instrument used to measure symptoms of generalised anxiety in the past 2 weeks. Similar to depression, anxiety and low mood are recognised as stress symptoms. Hence, measuring anxiety symptoms will aid with identifying stress levels. Examples of the item are "Worrying too much about different things" and "Trouble relaxing". The same response scale as PHQ-9 is used, where higher scores reflect more symptoms. Similar to the PHQ-9, the internal reliability of GAD-7 is excellent with Cronbach's α = .92.
Change in coping self-efficacy | Baseline, 8 days (completion of intervention), 4 weeks (follow-up)
  Coping Self-Efficacy Scale (CSES; Chesney et al., 2006) is a 26-item self-report instrument used to measure perceived self-efficacy for coping with threats and challenges. The items include "Keep from feeling sad" and "Resist the impulse to act hastily when under pressure". A 11-point scale is used (0 = 'Cannot do at all'; 5 = 'Moderately certain can do'; 10 = 'Certain can do'). A higher score denotes greater belief in one's coping abilities. The CSE possesses an excellent internal consistency of Cronbach's α= 0.95.
Psychological mindedness | Baseline
  Psychological Mindedness Scale (PM; Conte et al., 1990) measures an individual's ability to reflect on psychological processes, emotional processing and interpersonal relationships. PM is a 45-item self-report instrument consisting of items such as "I often find myself thinking about what made me act in a certain way" and "I am sensitive to the changes in my own feelings". It utilises a 4-point scale to score items (4 = 'Strongly agree'; 1 = 'Strongly disagree'). Higher total scores indicate higher levels of psychological mindedness. The PM produced a good internal consistency of Cronbach's α= 0.86.

OTHER OUTCOMES:
Engagement with the mobile application | 8 days (completion of intervention)
  An App Engagement Scale (Bakker & Rickard, 2018) assesses the strength of app engagement which is included as a manipulation check. This scale is a 7-item measure using a 5-point Likert scale (1 = 'Strongly disagree'; 5 = 'Strongly agree'). The scale has good internal reliability where Cronbach's α = .83. App engagement is predictive of positive outcomes on measures of mood and anxiety (Bakker & Rickard, 2018); should group differences emerge, app engagement will be controlled for in the statistical comparisons.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Suendermann, Ph.D., Principal Investigator — National University of Singapore
Locations (1):
- National University of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bakker D, Rickard N. Engagement in mobile phone app for self-monitoring of emotional wellbeing predicts changes in mental health: MoodPrism. J Affect Disord. 2018 Feb;227:432-442. doi: 10.1016/j.jad.2017.11.016. Epub 2017 Nov 9. PMID 29154165
- [Background] Chesney MA, Neilands TB, Chambers DB, Taylor JM, Folkman S. A validity and reliability study of the coping self-efficacy scale. Br J Health Psychol. 2006 Sep;11(Pt 3):421-37. doi: 10.1348/135910705X53155. PMID 16870053
- [Background] Conte HR, Plutchik R, Jung BB, Picard S, Karasu TB, Lotterman A. Psychological mindedness as a predictor of psychotherapy outcome: a preliminary report. Compr Psychiatry. 1990 Sep-Oct;31(5):426-31. doi: 10.1016/0010-440x(90)90027-p. PMID 2225801
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Derived] Toh SHY, Tan JHY, Kosasih FR, Sundermann O. Efficacy of the Mental Health App Intellect to Reduce Stress: Randomized Controlled Trial With a 1-Month Follow-up. JMIR Form Res. 2022 Dec 14;6(12):e40723. doi: 10.2196/40723. PMID 36515984